CLINICAL TRIAL: NCT01035879
Title: Phase 2, Randomized, Double-Blind, Placebo and Active-Comparator Controlled Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of MBX-2982 Administered Daily for 4 Weeks as Monotherapy in Patients With Type 2 Diabetes
Brief Title: Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of MBX-2982 Administered Daily for 4 Weeks as Monotherapy in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M2982-20920
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — MBX-2982; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- MBX-2982 25 mg (Experimental)
  Interventions: Drug: MBX-2982
- MBX-2982 100 mg (Experimental)
  Interventions: Drug: MBX-2982
- MBX-2982 300 mg (Experimental)
  Interventions: Drug: MBX-2982
- Sitagliptin 100 mg (Active Comparator)
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: MBX-2982 — tablets and capsule once daily
  Arms: MBX-2982 25 mg
Drug: MBX-2982 — tablets and capsule once daily
  Arms: MBX-2982 100 mg
Drug: MBX-2982 — tablets and capsule once daily
  Arms: MBX-2982 300 mg
Drug: Sitagliptin — tablets and capsule once daily
  Arms: Sitagliptin 100 mg
Drug: placebo — tablets and capsule once daily
  Arms: Placebo

SUMMARY:
To define the relative efficacy, safety and tolerability profiles of oral daily MBX-2982 at three different daily doses vs. placebo and sitagliptin 100 mg when administered for up to 4 weeks in patients that are treatment-naive or taking a single anti-diabetic medication (non-TZD, non-injectable).

DETAILED DESCRIPTION:
Approximately 100 patients will be randomized in this study, 20 to each of of the three MBX-2982 treatment groups, 20 to placebo, and 20 to the sitagliptin group. Patients will be taking 3 tablets and 1 capsule daily. This sample size provides the minimum number expected to ensure a power of at least 80% to detect a 20% decrease in the weighted mean glucose level associated with an extended mixed meal tolerance test (with 2 standardized meals) relative to placebo after 4 weeks of daily treatment with MBX-2982, assuming a drop-out rate of 20% and a common SD of 25%.

ELIGIBILITY:
Inclusion Criteria:

* History of type 2 diabetes of at least 3 months duration
* Treatment-naïve (not on any anti-diabetic medication) or treated with a single anti-diabetic agent (excluding insulin, exenatide or other GLP-1 analogs, pioglitazone or rosiglitazone)
* HbA1c 7.0-8.5% (inclusive) at screening
* BMI ≥ 26 kg/m2 for patients recruited from U.S or Georgia or ≥ 22 kg/m2 for patients recruited from India

Exclusion Criteria:

* Any history of type 1 diabetes or diabetic ketoacidosis
* History of major upper GI surgery
* Evidence or history of clinically significant GI illness including dyspepsia, PUD, nausea, diarrhea, malabsorption, etc.
* History of outpatient insulin use within last 1 year (insulin use while hospitalized is acceptable)
* Weight loss > 10 pounds (4.5 kg) in the 3 months prior to screening visit or use of weight loss medications (prescription or OTC) within 30 days of screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of MBX-2982 on the absolute and percent change from baseline and placebo in mean weighted average of 14-point blood glucose levels associated with a standardized breakfast and lunch | 4 weeks

SECONDARY OUTCOMES:
Evaluate the effect of MBX-2982 on additional glycemic parameters. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian Roberts, MD, Study Director — Metabolex, Inc.
Locations (14):
- United States (4):
  - Impact Clinical Trials, Los Angeles, California
  - Nevada Alliance Against Diabetes, Las Vegas, Nevada
  - United Medical Associates, Binghamton, New York
  - dgd Research, Inc., a Cetero Research Co., San Antonio, Texas
- Georgia (3):
  - Healthy Life Clinical Diagnostic Center, Tbilisi
  - Georgian Diabetes Center, Tbilisi
  - Medulla Chemotherapy and Immunotherapy Clinic, Tbilisi
- India (7):
  - Bharti Research Institute of Diabetes and Endocrinology, Karnāl, Haryana
  - Diabetes Thyroid Hormone Research Institute Pvt Ltd, Indore, M.p.
  - Gandhi Endocrinology & Diabetes Centre, Rāmdaspeth, Nagpur
  - Gokula Metropolis Research, MS Ramaiah Memorial Hospital, Bangalore
  - Medisys Clinisearch India Pvt Ltd, Bangalore
  - Hormone Care Research Centre, Ghaziabad
  - Bangalore Endocrinology & Diabetes Research Centre, Malleshwaram